CLINICAL TRIAL: NCT02904187
Title: Cerebral Activation and Bilateral Stimulation by Cochlear Implantation in Bilateral Deaf Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2008-542
Record Dates: First submitted 2016-08-11; First posted 2016-09-16 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Profound deaf patients (Other): Profound deaf patients with bilateral cochlear implants: Cortical brain activation pattern obtained by PET and EEG
  Interventions: Other: Positron Emission Tomography (PET); Other: Electroencephalogram (EEG)
- Healthy volunteers (Other): Healthy volunteers: Cortical brain activation pattern obtained by PET and EEG
  Interventions: Other: Positron Emission Tomography (PET); Other: Electroencephalogram (EEG)

INTERVENTIONS:
Other: Positron Emission Tomography (PET)
Other: Electroencephalogram (EEG)

SUMMARY:
The primary objective to this study is to describe bilateral auditory information processing in profoundly deaf patients with bilateral cochlear implants compared with normal hearing patients. Assumption used is that due to the central consequences of bilateral deafness on binaural auditory information central processing, time between activation of the two cochlear implants is a decisive factor in bilateral implantation compared to unilateral implantation

ELIGIBILITY:
Inclusion criteria for patients:

- profoundly deaf patients with bilateral cochlear implants

Exclusion criteria for patients:

* post-operative complications
* incomplete surgical insertion of one of the cochlear implant
* age under 18 years
* non-compliant patient
* pregnant woman or woman with no efficient contraception method
* informed consent not signed
* no health insurance

Inclusion criteria for control

- normal hearing subjects

Exclusion criteria control

* normal hearing subject
* subject under 18 years old
* unilateral or bilateral hearing loss
* non-compliant subject
* pregnant woman or woman with no efficient contraception method
* informed consent not signed
* no health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-03-17 (Actual); Primary Completion 2016-03-22 (Actual); Study Completion 2016-03-22 (Actual)

PRIMARY OUTCOMES:
Cortical brain activation pattern | 6 months
  Cortical brain activation pattern obtained by PET or EEG cartography. Activation pattern will be compared between normal hearing subjects and deaf adults with bilateral cochlear implants

CONTACTS AND LOCATIONS:
Locations (1):
- Département d'ORL, Hôpital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coudert A, Verdelet G, Reilly KT, Truy E, Gaveau V. Intensive Training of Spatial Hearing Promotes Auditory Abilities of Bilateral Cochlear Implant Adults: A Pilot Study. Ear Hear. 2023 Jan-Feb 01;44(1):61-76. doi: 10.1097/AUD.0000000000001256. Epub 2022 Aug 9. PMID 35943235